CLINICAL TRIAL: NCT02781545
Title: Predicting and Monitoring Motor Development of Children Requiring Surgery as Neonates for Complex Congenital Heart Disease
Brief Title: Motor Development of Children That Have Surgery as Newborns for Complex Congenital Heart Disease
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Advocate Center for Pediatric Research (Other); University Medical Center Groningen (Other)
Responsible Party: Sponsor
Other Study IDs: AHC IRB#6036
Record Dates: First submitted 2016-05-18; First posted 2016-05-24 (Estimated); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Heart Defects, Congenital
Keywords: Child Development; Psychomotor Performance; Newborns; Surgery
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Infants requiring surgery in the neonatal period for complex congenital heart diseases are at risk for developmental problems. For infants with congenital heart diseases with admixture physiology and single ventricles, optimal circulation is associated with signs of adequate systemic perfusion and a systemic arterial oxygen saturation typically between 75% to 90%. Infants are often unable to withstand standardized developmental testing during early infancy due to medical fragility and sternal precautions after surgery. Evaluation of the quality of spontaneous movements and movement variability is a good alternative. The quality of general movements in early infancy is a valid predictor of neurological disorders in high risk infant groups and is assessed with short periods of video-recorded observations. This methodology has yet to be studied in infants with complex congenital heart disease that require surgery as neonates. For older infants, the Infant Motor Profile (IMP) is a promising tool to document developmental outcome.

DETAILED DESCRIPTION:
Congenital heart defects (CHD) are conditions present at birth and affect heart structure, function, and manner in which blood flows through the heart and to the rest of the body. The incidence of severe CHD is about 2.5 to 3/1,000 live births. With improvements in cardiac surgical technique and critical care medicine, the vast majority of babies with CHD are expected to survive to school age and beyond. However, these surgical and medical advances are also associated with increased risk for neurodevelopmental morbidity.

Traditionally, a quantitative approach measured gross motor development of infants at risk for delay, including children with complex congenital heart disease. These tools emphasize elicited responses; however, clinical use and validity may be limited by the infant's behavioral state, unstable physiological status, intolerance of handling, or sternal/surgical precautions. Alternatively, European clinicians working in the field of developmental neurology realized that variation and adaptability in motor behavior may assist in the evaluation of motor development. The application of motor variation and adaptability as a means to evaluate neuromotor condition in early infancy was significant for early detection of infants at high risk for developmental problems or cerebral palsy in a number of studies with high-risk infant groups. This form of evaluation has yet to be studied in infants with complex congenital heart diseases.

The proposed study aims to study motor development of two infant groups based on oxygen saturation targets after neonatal surgery and to study the validity of the assessment tools based on the quality of movement variation and adaptability, i.e., the General Movements Assessment (GMsA) and the Infant Motor Profile (IMP) in infants with complex congenital heart disease.

Hypothesis:

Baseline oxygen saturation after neonatal heart surgery in children with complex congenital heart diseases is a determinant of motor performance outcome at 18 months on the Infant Motor Profile.

Specific Objectives:

1. To determine developmental outcomes at 18 months in two infant groups based on oxygen saturation targets.
2. To validate specific neuromotor assessment tools that determine developmental outcome in two infant groups based on oxygen saturation targets.

Specific Aims:

1. To compare motor outcomes at 18 months measured with the IMP of two groups of infants who had surgery as neonates for complex congenital heart disease grouped by baseline oxygen saturation targets after the first surgery (≥ 90%; high saturation and < 90%; low saturation, i.e., admixed lesions).
2. To describe the quality of general movements from birth through three months at five assessment points in infants with high oxygen saturation and infants with low oxygen saturation.
3. To describe motor development in terms of IMP-scores at 6, 12 and 18 months in infants with high oxygen saturation and infants with low oxygen saturation.
4. To explore the predictive value of GMsA at three months in a pooled group of infants with high oxygen saturation and low oxygen saturation with development outcome at 18 months assessed with:

   1. Infant Motor Profile (IMP)
   2. Alberta Infant Motor Scales (AIMS)
   3. Motor Composite score of the Bayley Scales of Infant Development, 3rd edition (BSID-3)
   4. Cognitive and Language composite scores of the BSID-3.
5. To determine the concurrent validity of the Infant Motor Profile (IMP) on the basis of comparison with:

   1. Alberta Infant Motor Scales (AIMS) at 6, 12, and 18 months.
   2. Bayley Motor Composite score at 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Infants diagnosed with complex congenital heart diseases that require surgery during the neonatal period, ages 0-30 days
* Surgical care at Advocate Christ Medical Center/Advocate Children's Hospital, Oak Lawn, Il

Exclusion Criteria:

* Chromosomal abnormalities and/or known syndromes

Max Age: 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Consecutive infant sampling of infants with complex congenital heart diseases
Sampling Method: Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2015-05; Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Motor development at 18 months | 18 months
  Comparison of motor development of two groups of infants based on oxygen saturation targets after neonatal surgery using the Infant Motor Profile

SECONDARY OUTCOMES:
Movement quality from birth to 4 months of age | 4 months. The infant's general movements are video-recorded three to five times from birth to four month according to this schedule: pre-operation (if possible), hospital discharge, one month of age, two months of age, and three months of age
  Comparison of the trajectory of movement quality for two infant groups based on video recorded General Movements Assessments for at least three assessment points from birth to 4 months of age
Concurrent validity | 18 months
  Assess concurrent validity of the Infant Motor Profile total score and performance score with the Alberta Infant Motor Scales at 6, 12, and 18 months, and the Bayley Scales of Infant Development (3rd edition) motor composite score at 18 months
Cognitive and language development at 18 months | 18 months
  Comparison of the two infant groups based on the cognitive and language composite scores of the Bayley Scales of Infant Development (3rd edition)

CONTACTS AND LOCATIONS:
Overall Officials: Darlene Huisenga, PT, DPT, PCS, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Advocate Children's Hospital, Oak Lawn, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Manuscript, Poster presentation, Conference presentation
Time Frame: 6 months after publication

REFERENCES:
- [Background] Donofrio MT, Duplessis AJ, Limperopoulos C. Impact of congenital heart disease on fetal brain development and injury. Curr Opin Pediatr. 2011 Oct;23(5):502-11. doi: 10.1097/MOP.0b013e32834aa583. PMID 21881507
- [Background] Hoffman JI, Kaplan S. The incidence of congenital heart disease. J Am Coll Cardiol. 2002 Jun 19;39(12):1890-900. doi: 10.1016/s0735-1097(02)01886-7. PMID 12084585
- [Background] Brosig CL, Mussatto KA, Kuhn EM, Tweddell JS. Neurodevelopmental outcome in preschool survivors of complex congenital heart disease: implications for clinical practice. J Pediatr Health Care. 2007 Jan-Feb;21(1):3-12. doi: 10.1016/j.pedhc.2006.03.008. PMID 17198894
- [Background] Limperopoulos C, Majnemer A, Shevell MI, Rosenblatt B, Rohlicek C, Tchervenkov C. Neurodevelopmental status of newborns and infants with congenital heart defects before and after open heart surgery. J Pediatr. 2000 Nov;137(5):638-45. doi: 10.1067/mpd.2000.109152. PMID 11060529
- [Background] Hadders-Algra M. Variation and variability: key words in human motor development. Phys Ther. 2010 Dec;90(12):1823-37. doi: 10.2522/ptj.20100006. Epub 2010 Oct 21. PMID 20966209
- [Background] Hadders-Algra M. General movements: A window for early identification of children at high risk for developmental disorders. J Pediatr. 2004 Aug;145(2 Suppl):S12-8. doi: 10.1016/j.jpeds.2004.05.017. PMID 15292882
- [Background] Hamer EG, Bos AF, Hadders-Algra M. Assessment of specific characteristics of abnormal general movements: does it enhance the prediction of cerebral palsy? Dev Med Child Neurol. 2011 Aug;53(8):751-6. doi: 10.1111/j.1469-8749.2011.04007.x. Epub 2011 Jun 29. PMID 21711457